CLINICAL TRIAL: NCT06833671
Title: Effect of Preoperative Two Hours Carbohydrate Load On Pediatric Patient Undergoing Elective Surgery: A Randomized Controlled Study
Brief Title: Preoperative Two Hours Carbohydrate Load On Pediatric Patient Undergoing Elective Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Amany Mohamed Abotaleb, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 35506/5/22
Record Dates: First submitted 2025-02-13; First posted 2025-02-19 (Actual); Last update posted 2025-02-19 (Actual); Status verified 2025-02

CONDITIONS: Preoperative; Carbohydrate; Pediatric; Elective Surgery
MeSH Terms: interventions — Glucose; Water

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Apple juice group (Experimental): A preoperative carbohydrate load was done two hours before the operation using a10 ml/kg, with a maximal volume of 250 ml of commercial brand of apple juice (glucose 28 g in 250 ml).
  Interventions: Other: Apple juice
- Anhydrous glucose group (Experimental): A preoperative carbohydrate load was done using 1.75mg/kg/dose of anhydrous glucose (Alpha Chmika).
  Interventions: Drug: Anhydrous glucose
- Water group (Other): Patients received water
  Interventions: Other: Water

INTERVENTIONS:
Other: Apple juice — A preoperative carbohydrate load was done two hours before the operation using a10 ml/kg, with a maximal volume of 250 ml of commercial brand of apple juice (glucose 28 g in 250 ml).
  Arms: Apple juice group
Drug: Anhydrous glucose — A preoperative carbohydrate load was done using 1.75mg/kg/dose of anhydrous glucose (Alpha Chmika).
  Arms: Anhydrous glucose group
Other: Water — Patients received water.
  Arms: Water group

SUMMARY:
This work evaluated the systemic effect of different preoperative carbohydrate (CHO) loads in pediatrics undergoing elective surgery.

DETAILED DESCRIPTION:
Children undergoing surgery experience stress due to disruptions in their daily routine and exposure to various perioperative circumstances that induce anxiety and pain.

The management of perioperative nutrition in pediatric patients is a crucial aspect of patient care.

The concept of preoperative carbohydrate (CHO) loading has gained attention as a potential strategy to mitigate these drawbacks. The administration of a CHO-rich drink two hours preoperative has been proposed to maintain euglycemia, decline IR, and enhance postoperative recovery

ELIGIBILITY:
Inclusion Criteria:

* Age from 5 to 10 years.
* Both sexes.
* American Society of Anesthesiologists (ASA) physical status I and II.
* Scheduled for elective surgery.

Exclusion Criteria:

* Diabetes mellitus.
* Insulin resistance (IR).
* Renal or hepatic insufficiency.
* Esophageal or gastric surgery or gastrointestinal disorders history (including gastroesophageal reflux, hiatal hernia, or gastritis).

Ages: 5 Years to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2024-10-21 (Actual); Study Completion 2024-10-21 (Actual)

PRIMARY OUTCOMES:
C-reactive protein (CRP) level | 4 hours postoperatively
  C-reactive protein (CRP) level was assessed two h before surgery as baseline, at induction of anesthesia, and 4 hours after the operation.

SECONDARY OUTCOMES:
Neutrophil/ lymphocyte ratio | 4 hours postoperatively
  Neutrophil/ lymphocyte ratio (NLR) was assessed 2 h before surgery as baseline, at induction of anesthesia, and 4 hours after the operation.
Level of procalcitonin | 4 hours postoperatively
  Level of procalcitonin was assessed two h before surgery as baseline, at induction of anesthesia, and 4 hours after the operation.
Homeostatic model assessment for insulin resistance | 4 hours postoperatively
  Homeostatic model assessment for insulin resistance(HOMA.IR) was assessed two h before surgery as baseline, at induction of anesthesia, and 4 hours after the operation.
Level of C-peptide | 4 hours postoperatively
  Level of C-peptide was assessed two h before surgery as baseline, at induction of anesthesia, and 4 hours after the operation.
Level of random blood glucose | Two hours before the surgery
  Level of random blood glucose (RBG) was measured at two hours before the surgery.
Patient's parent's satisfaction | 4 hours postoperatively
  Parent satisfaction level was evaluated by 3-point Likert scale (1, unsatisfied; 2, neutral; 3, satisfied).
Incidence of complications | 4 hours postoperatively
  Incidence of complications such as perioperative nausea, vomiting, and aspiration were documented.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, El-Gharbia, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.

REFERENCES:
- [Derived] Abdelwahed WMA, Abdelelsalam WM, Taha OA, Abdelbadie S, Taleb AMA. Effect of Preoperative 2-Hour Carbohydrate Load on Pediatric Patients Undergoing Elective Surgery: A Randomized Controlled Study. Anesthesiol Res Pract. 2025 Dec 3;2025:5580879. doi: 10.1155/anrp/5580879. eCollection 2025. PMID 41357678